CLINICAL TRIAL: NCT01901393
Title: A Multicenter, Prospective, Randomized, Double-blind Study to Determine the Efficacy of Intravenous Ibuprofen Compared to Intravenous Ketorolac for Pain Control Following Arthroscopic Knee Surgery
Brief Title: Efficacy of Intravenous Ibuprofen Compared to Intravenous Ketorolac for Pain Control Following Arthroscopic Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-CL-020
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: Post Operative Pain,; Pail relief
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Ibuprofen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV ibuprofen (Experimental): 800mg ibuprofen
  Interventions: Drug: IV ibuprofen
- ketorolac (Active Comparator): 30mg ketorolac
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: IV ibuprofen
  Other Names: Caldolor
  Arms: IV ibuprofen
Drug: Ketorolac
  Other Names: Ketorolac Tromethamine
  Arms: ketorolac

SUMMARY:
The purpose of this study is to assess the efficacy of intravenous ibuprofen compared to ketorolac for the treatment of postoperative pain as measured by patient pain intensity (Visual Analog Scale, VAS)

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for knee arthroscopy

Exclusion Criteria:

* Inadequate IV access.
* History of allergy or hypersensitivity to any component of ibuprofen, ketorolac, aspirin (or aspirin related products), non-steroidal anti-inflammatory drugs (NSAIDs), opioids or cyclooxygenase-2 (COX-2) inhibitors.
* Less than 18 years of age.
* Use of analgesics less than 8 hours prior to surgery.
* Patients with active, clinically significant anemia.
* History or evidence of asthma or heart failure.
* Pregnant.
* Recent history of chronic opioid use.
* Concomitant use of probenecid.
* Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions and to return for the required assessments.
* Refusal to provide written authorization for use and disclosure of protected health information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur P Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - Rush University Medical Center, Chicago, Illinois
  - North Mississippi Sports Medicine & Orthopaedic Clinic, Tupelo, Mississippi
  - The Ohio State University Vexner Medical Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Ibuprofen: 800mg ibuprofen
  IV ibuprofen
- Ketorolac: 30mg ketorolac
  Ketorolac
Period: Overall Study
Arm/Group | IV Ibuprofen | Ketorolac
Started | 51 | 49
Completed | 50 | 49
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat population consisted of all subjects who were enrolled and received at least a partial dose of investigational medicinal product.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Ibuprofen | Ketorolac | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13.3) | 46 (15.5) | 46 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 33 | 28 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 49 | 47 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 44 | 48 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pain Relief (Pain Intensity at Rest)
Description: Pain assessed using VAS (Visual Analog Scale, VAS). The VAS is a continuous scale compromised of a horizontal line, one hundred millimeters in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between 0 (No Pain) and 100 (Worst Possible Pain).
Time Frame: First possible time post-surgery, an expected average of 6 hours
Population: This analysis was performed on all subject who completed the VAS at Rest Immediately Following their Procedure
Measure: Mean (Standard Deviation); unit: units on a scale (in mm)
Arm/Group | IV Ibuprofen | Ketorolac
Number analyzed (Participants) | 50 | 49
units on a scale (in mm) | 30 (27.0) | 32 (25.1)

2. Secondary Outcome: Rescue Medication Use in Post-operative Period
Description: Amount of rescue medication (in milligrams) will be measured
Time Frame: Post-operative period until discharge, an expected average of 6 hours
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | IV Ibuprofen | Ketorolac
Number analyzed (Participants) | 51 | 49
milligrams
  Narcotic | 13.7 (17.19) | 13.2 (16.50)
  Acetaminophen | 188.5 (255.06) | 179.1 (248.77)

3. Secondary Outcome: Time to First Use of Rescue Med Will be Measured
Description: Time to first rescue medication (in hours) in the postoperative period through discharge.
Time Frame: Post-operative period until discharge, an expected average of 6 hours
Measure: Mean (Standard Error); unit: hours
Arm/Group | IV Ibuprofen | Ketorolac
Number analyzed (Participants) | 51 | 49
hours | 1.2 (0.11) | 1.2 (0.10)

4. Secondary Outcome: Patient Satisfaction
Description: Measured using 2 question, 4 point scale.
Time Frame: Post-operative period until discharge, an expected average of 6 hours
Measure: Number; unit: Participants
Arm/Group | IV Ibuprofen | Ketorolac
Number analyzed (Participants) | 51 | 49
Participants
  Poor | 0 | 1
  Fair | 4 | 8
  Good | 20 | 18
  Excellent | 26 | 22

5. Secondary Outcome: Incidence of Serious Adverse Events
Description: Number of subjects experiencing treatment-emergent serious adverse events
Time Frame: Post-operative period until discharge, an expected average of 6 hours
Measure: Number; unit: Number of events
Arm/Group | IV Ibuprofen | Ketorolac
Number analyzed (Participants) | 51 | 49
Number of events | 0 | 0

6. Primary Outcome: Efficacy of Pain Relief (Pain Intensity With Movement)
Description: as for outcome 1
Time Frame: First possible time post-surgery, an expected average of 6 hours
Population: This analysis was performed on all subject who completed the VAS with Movement Immediately Following their Procedure
Measure: Mean (Standard Deviation); unit: units on a scale (in mm)
Arm/Group | IV Ibuprofen | Ketorolac
Number analyzed (Participants) | 49 | 47
units on a scale (in mm) | 32 (28.0) | 41 (28.2)

ADVERSE EVENTS:
Arm/Group | IV Ibuprofen | Ketorolac
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 0/51 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No